CLINICAL TRIAL: NCT05127044
Title: Characterization of Pre-Term Neonatal Skin by Diffuse Reflectance Spectroscopy Pilot Study
Brief Title: Characterization of Pre-Term Neonatal Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 263337
Record Dates: First submitted 2021-10-14; First posted 2021-11-19 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: Skin Disorder
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Qualified Preterm Infants (Other): The skin of preterm neonates will be analyzed with diffuse reflectance spectroscopy (DRS) and Philip's BiliChek transcutaneous bilirubin testing for baseline comparison
  Interventions: Device: Diffuse Reflectance Spectroscopy; Diagnostic Test: BiliChek

INTERVENTIONS:
Device: Diffuse Reflectance Spectroscopy — DRS will be used as a non-invasive optical spectroscopy method to evaluate whether DRS spectra can be used to extract optical information related to skin maturity as well as hemoglobin, melanin, and bilirubin concentrations.
  Other Names: DRS
Diagnostic Test: BiliChek — BiliChek will be used as a control for determining bilirubin content.
  Other Names: Transcutaneous Bilirubin Reading

SUMMARY:
The skin of pre-term neonates is not fully developed and often leads to trans-epidermal water loss, trouble regulating temperature, and increased risk of skin wounds. Current treatment decisions are based on subjective, qualitative assessments of the skin. The purpose of this pilot study is to evaluate the utility of non-invasive optical spectroscopy methods to collect key biological information from neonatal skin, including skin maturity, blood oxygenation, and bilirubin content. Parents of pre-term neonatal subjects (n=44) will be recruited for consent to participate, and spectral measurements will be made with a diffuse reflectance spectrometer(DRS) device previously approved by the University of Arkansas for Medical Sciences Institutional Review Board. The spectral data will be analyzed to extract parameters related to tissue light scattering, oxy-and deoxy-hemoglobin, melanin, and bilirubin. The system will be validated by comparing extracted spectra with expected literature values and directly correlating the measured bilirubin levels with readouts from the current University of Arkansas for Medical Sciences practice standard: Philip's BiliChek. The long-term goal is to develop and use non-invasive optical readouts to predict and monitor skin dysfunction in the Neonatal Intensive Care Unit (NICU).

DETAILED DESCRIPTION:
This is a cross-sectional, pilot study to characterize the response of neonatal premature skin to DRS when excited with a white light source, and provide a baseline of how the collected spectra change with the maturation of the epidermal layer in the weeks to term gestation after birth. DRS spectra and BiliChek measurements will be performed on the study population admitted to the Neonatal Intensive Care Unit. The pilot data will be used to evaluate whether Diffuse Reflectance Spectroscopy spectra can be used to extract optical information on skin maturity as well as hemoglobin, melanin, and bilirubin concentrations. The investigators will extract spectra for each chromophore and the relative concentration from the Diffuse Reflectance Spectroscopy measurements. Extracted Diffuse Reflectance Spectroscopy spectra will be compared to published absorbance spectra for each chromophore. The criteria for success will be a high, positive correlation (r ≥ 0.85) between the extracted Diffuse Reflectance Spectroscopy bilirubin concentration and BiliChek-derived concentration.

The following coded data will also be collected to investigate correlations with the Diffuse Reflectance Spectroscopy spectra: blood oxygen saturation, weight, ethnicity, corrected age, gestational age, sex, most recent complete blood count (if available, or partial count if not), most recent chemistry levels, lipids, liver profile, and blood gas (all if available). BiliChek measurements of bilirubin content will be compared to the extracted bilirubin contribution measured from the Diffuse Reflectance Spectroscopy spectra using linear regression and assessed using Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than or equal to 37 weeks gestation at birth
* Current care provided by the UAMS NICU

Exclusion Criteria:

* Infants entering palliative care
* Infants with known liver disease
* Infants on isolation precautions
* Infants at end of life
* On minimal stimulation protocol
* Any other condition, that in the opinion of the investigator, might interfere with the safe conduct of the study or place the subject at increased risk

Ages: 24 Hours to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sartini, DNP, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacques, S.L., D.G. Oelberg, and I. Saidi, Method and apparatus for optical measurement of bilirubin in tissue. 1994, Board of Regents, The University of Texas System: United States.
- [Result] Afsar FS. Physiological skin conditions of preterm and term neonates. Clin Exp Dermatol. 2010 Jun;35(4):346-50. doi: 10.1111/j.1365-2230.2009.03562.x. Epub 2009 Sep 15. PMID 19758381
- [Result] Zonios G, Bykowski J, Kollias N. Skin melanin, hemoglobin, and light scattering properties can be quantitatively assessed in vivo using diffuse reflectance spectroscopy. J Invest Dermatol. 2001 Dec;117(6):1452-7. doi: 10.1046/j.0022-202x.2001.01577.x. PMID 11886508
- [Result] Subhash N, Mallia JR, Thomas SS, Mathews A, Sebastian P, Madhavan J. Oral cancer detection using diffuse reflectance spectral ratio R540/R575 of oxygenated hemoglobin bands. J Biomed Opt. 2006 Jan-Feb;11(1):014018. doi: 10.1117/1.2165184. PMID 16526895
- [Result] Qualter YM, Allen NM, Corcoran JD, O'Donovan DJ. Transcutaneous bilirubin--comparing the accuracy of BiliChek(R) and JM 103(R) in a regional postnatal unit. J Matern Fetal Neonatal Med. 2011 Feb;24(2):267-70. doi: 10.3109/14767058.2010.484471. Epub 2010 May 19. PMID 20482289
- [Result] Rajaram N, Nguyen TH, Tunnell JW. Lookup table-based inverse model for determining optical properties of turbid media. J Biomed Opt. 2008 Sep-Oct;13(5):050501. doi: 10.1117/1.2981797. PMID 19021373

RESULTS

PARTICIPANT FLOW:
Groups:
- Qualified Preterm Infants: Preterm infants will receive non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS will be used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin including skin maturity, blood oxygenation, and bilirubin content.
  BiliChek: BiliChek will be used as a control for determining bilirubin content.
Period: Overall Study
Arm/Group | Qualified Preterm Infants
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Qualified Preterm Infants
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Gestational Age in Weeks] | 33.3 [23 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Qualified Preterm Infants
  participants
    United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Bilirubin Concentration From Non-invasive Diffuse Reflectance Spectroscopy (DRS) vs BiliChek
Description: Number of participants with premature skin assessed with Diffuse Reflectance Spectroscopy, comparing bilirubin concentration levels/readings produced by DRS system with readouts from the current UAMS practice standard (Philip's BiliChek) using a linear regression and a Pearson's correlation coefficient assessment.
Time Frame: 15 Minutes
Population: All infants received the same testing method on each area of infant body
Measure: Number; unit: Correlation Coefficient R-Value
Groups:
- Qualified Preterm Infants-Chest: Preterm infants received non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin: Chest
  BiliChek: BiliChek will be used as a control for determining bilirubin content.
- Qualified Preterm Infants-Upper Arm: Preterm infants received non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin: Upper Arm
  BiliChek: BiliChek will be used as a control for determining bilirubin content.
- Qualified Preterm Infants-Outer Thigh: Preterm infants received non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin: Outer Thigh
  BiliChek: BiliChek will be used as a control for determining bilirubin content.
- Qualified Preterm Infants- Forehead: Preterm infants received non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin: Forehead
  BiliChek: BiliChek will be used as a control for determining bilirubin content.
- Qualified Preterm Infant- Subject Mean: Preterm infants received non-invasive optical spectroscopy and transcutaneous bilirubin testing for baseline comparison
  Diffuse Reflectance Spectroscopy: DRS used as a non-invasive optical spectroscopy method to collect key biological information from neonatal skin: Mean Analysis
  BiliChek: BiliChek will be used as a control for determining bilirubin content
Arm/Group | Qualified Preterm Infants-Chest | Qualified Preterm Infants-Upper Arm | Qualified Preterm Infants-Outer Thigh | Qualified Preterm Infants- Forehead | Qualified Preterm Infant- Subject Mean
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
Correlation Coefficient R-Value | 0.814386451 | 0.85422779 | 0.67588721 | 0.79293382 | 0.86294585
Statistical Analysis 1: Comparison: Qualified Preterm Infants-Chest; Power calculation located in Study Protocol-Correlation Coefficient-R Value; Test type: Other — An a priori power analysis was conducted to determine the number of subjects needed to detect a similar strong correlation between the DRS and BiliChek data (α = 0.05, power = 0.8, r0 = 0.7, r1 = 0,85; G*Power3.1). For this study n = 44 subjects (from Study Protocol); Multiple R = 0.81438645
Statistical Analysis 2: Comparison: Qualified Preterm Infants-Upper Arm; Power calculation located in Study Protocol; Test type: Other — [test comment as in outcome 1, analysis 1]; Multiple R = 0.85442277
Statistical Analysis 3: Comparison: Qualified Preterm Infants-Outer Thigh; Power calculation located in Study Protocol; Test type: Other — [test comment as in outcome 1, analysis 1]; Multiple R = 0.0758872
Statistical Analysis 4: Comparison: Qualified Preterm Infants- Forehead; Power calculation located in Study Protocol; Test type: Other — [test comment as in outcome 1, analysis 1]; Multiple R = 0.7929338
Statistical Analysis 5: Comparison: Qualified Preterm Infant- Subject Mean; Power calculation located in Study Protocol; Test type: Other — [test comment as in outcome 1, analysis 1]; Multiple R = 0.86294585

2. Secondary Outcome: Hemoglobin Readings From Diffuse Reflectance Spectroscopy (DRS) Spectra Compared With Expected Values
Description: Compare hemoglobin readings from the DRS system's extracted spectra with expected values by gestational age, race, ethnicity, and sex using a linear regression and a Pearson's correlation coefficient assessment.
Time Frame: approximately one day per subject
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Qualified Preterm Infants
Number analyzed (Participants) | 44
g/L | 6.03 (0.843)
Statistical Analysis 1: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between hemoglobin concentration and weight; p = 0.1544, Linear correlation; Pearson Correlation Coefficient = -0.2184
Statistical Analysis 2: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between hemoglobin concentration and gestational age; p = 0.0087, Linear correlation; Pearson Correlation Coefficient = 0.3909
Statistical Analysis 3: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with hemoglobin concentration as the dependent variable and sex as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.3038, Regression, Linear; Coefficient of determination = 0.0252
Statistical Analysis 4: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with hemoglobin concentration as the dependent variable and ethnicity as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.6434, Regression, Linear; Coefficient of determination = 0.0213
Statistical Analysis 5: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with hemoglobin concentration as the dependent variable and weight as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.1544, Regression, Linear; Coefficient of determination = 0.0477
Statistical Analysis 6: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with hemoglobin concentration as the dependent variable and gestational age as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.0087, Regression, Linear; Coefficient of determination = 0.1528

3. Secondary Outcome: Melanin Readings From Diffuse Reflectance Spectroscopy (DRS) Spectra Compared With Expected Values
Description: Compare melanin readings from the DRS system's extracted spectra with expected values by gestational age, race, ethnicity, and sex using a linear regression and a Pearson's correlation coefficient assessment.
Time Frame: approximately one day per subject
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Qualified Preterm Infants
Number analyzed (Participants) | 44
mg/dL | 3.19 (1.24)
Statistical Analysis 1: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between melanin concentration and weight; p = 0.3143, Linear correlation; Pearson Correlation Coefficient = -0.1552
Statistical Analysis 2: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between melanin concentration and gestational age; p = 0.5914, Linear correlation; Pearson Correlation Coefficient = -0.0832
Statistical Analysis 3: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with melanin concentration as the dependent variable and sex as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.868, Regression, Linear; Coefficient of determination = 0.000665
Statistical Analysis 4: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with melanin concentration as the dependent variable and ethnicity as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.0001, Regression, Linear; Coefficient of determination = 0.574
Statistical Analysis 5: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with melanin concentration as the dependent variable and weight as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.3143, Regression, Linear; Coefficient of determination = 0.0241
Statistical Analysis 6: Comparison: Qualified Preterm Infants; Test type: Other — A simple linear regression model was fitted with melanin concentration as the dependent variable and gestational age as the independent predictor. The strength of the relationship was evaluated using the coefficient of determination (R²); p = 0.5914, Regression, Linear; Coefficient of determination = 0.0069

4. Secondary Outcome: Bilirubin Readings From Diffuse Reflectance Spectroscopy (DRS) Spectra Compared With Expected Values
Description: Compare bilirubin readings from the DRS system's extracted spectra with expected values by gestational age, race, ethnicity, and sex using a linear regression and a Pearson's correlation coefficient assessment.
Time Frame: approximately one day per subject
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Qualified Preterm Infants
Number analyzed (Participants) | 44
mg/dL | 7.34 (3.91)
Statistical Analysis 1: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between bilirubin concentration and weight; p = 0.8203, Linear correlation; Pearson Correlation Coefficient = -0.0353
Statistical Analysis 2: Comparison: Qualified Preterm Infants; Test type: Other — Pearson's correlation coefficient was calculated to assess the relationship between bilirubin concentration and gestational age; p = 0.0001, Linear correlation; Pearson Correlation Coefficient = 0.595
Statistical Analysis 3: Comparison: Qualified Preterm Infants; Test type: Other — [test comment as in outcome 3, analysis 3]; p = 0.2156, Regression, Linear; Coefficient of determination = 0.0363
Statistical Analysis 4: Comparison: Qualified Preterm Infants; Test type: Other — [test comment as in outcome 3, analysis 4]; p = 0.0066, Regression, Linear; Coefficient of determination = 0.2172
Statistical Analysis 5: Comparison: Qualified Preterm Infants; Test type: Other — [test comment as in outcome 3, analysis 5]; p = 0.8203, Regression, Linear; Coefficient of determination = 0.00124
Statistical Analysis 6: Comparison: Qualified Preterm Infants; Test type: Other — [test comment as in outcome 3, analysis 6]; p = 0.0001, Regression, Linear; Coefficient of determination = 0.354

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Qualified Preterm Infants
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT05127044/Prot_SAP_000.pdf